CLINICAL TRIAL: NCT05276661
Title: Chia Nan University of Pharmacy & Science
Brief Title: A Project to Study Probiotic Beauty Products on Skin Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chia Nan University of Pharmacy ＆ Science (Other)
Collaborators: Glac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSMHIRB-2-R-025-2.1
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "A" gel (TAC/Collagen gel) (Experimental): The "A" gel (TAC/Collagen gel) was applied on subjects' right face
  Interventions: Dietary Supplement: TAC/Collagen gel
- "B" gel (placebo lotion) (Placebo Comparator): the "B" gel (placebo lotion) on their left face
  Interventions: Dietary Supplement: placebo lotion

INTERVENTIONS:
Dietary Supplement: TAC/Collagen gel — Apply it twice per day for 4 weeks
  Arms: "A" gel (TAC/Collagen gel)
Dietary Supplement: placebo lotion — Apply it twice per day for 4 weeks
  Arms: "B" gel (placebo lotion)

SUMMARY:
The aim of the study was to use probiotic beauty products for 4 weeks and evaluate the impact of products on healthy skin.

DETAILED DESCRIPTION:
Twenty subjects were recruited and informed to apply the lotion gel twice per day (3~5 mg/cm2 once) for 4 weeks. Two kinds of facial lotiongels, "A" gel and "B" gel, were provided to every subject. The "A" gel (TAC/Collagen lotiongel) was applied on subjects' right face and the "B" gel (placebo lotion) on their left face (formula showed as Table S2). Ordinary cosmetics usage was permitted but any change of usage was not allowed during the intervention. Outdoor activities (sun exposure) and the usage of sunscreen lotion were not limited in this study. Every subject was required to inspect his/her skin condition on week 0 and 4. Before inspection, the face was washed with water and waited for 30 min in an air-conditioned room (25°C, humility 55 ± 5%). Among these 20 subjects, eight of them had severe acne with at least two acne lesions on each side of face when participating this trial. They were instructed for more visits to evaluate the symptom of acne on week 1 and 2.

Skin hydration (Corneometer CM825, Courage + Khazaka Electroni, Germany), sebum (Callegari 1930, Italy), and inflammation detection (Chroma Meter MM-500, Minolta, Japan) of upper cheek were measured in every subject. The improvement in inflammation was positively correlated with a decrease of a* value or an increase of L* value. VISIA® Complexion Analysis (VISIA® Complexion Analysis, U.S.A.) was also employed to measure the skin inflammation, porphyrins numbers and brown spot numbers of whole face. The result was presented as the mean value and the relative percentage (%) to the baseline.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers aged above 20 years old

Exclusion Criteria:

1. Subject with diseases of the skin, heart, liver, kidney, endocrine and other organs and patients with mental illness (according to medical history).
2. Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
3. Female who is pregnant or nursing or planning to become pregnant during the course of the study.
4. Received facial laser therapy, chemical peeling or UV overexposure in the past 4 weeks.
5. Involuntary subject
6. People who is taking chronic disease medication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Effects of the TAC/Collagen Gel on Human Skin Hydration | Subjects will be tested in the 4th week
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
Effects of the TAC/Collagen Gel on Human Skin Sebum | Subjects will be tested in the 4th week
  Callegari 1930 was utilized to measure skin inflammation. Units: arbitrary units.
Effects of the TAC/Collagen gel on Human Skin Inflammation | Subjects will be tested in the 4th week
  Chroma Meter MM-500 was utilized to measure skin inflammation. Units: arbitrary units.
Effect of TAC/Collagen Gel on Human Acne Healing and Porphyrins Numbers | Subjects will be tested in the 4th week
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
Effects of the TAC/Collagen Gel on Human Skin Brown Spot Numbers | Subjects will be tested in the 4th week
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, PhD, Principal Investigator — Chia Nan University of Pharmacy ＆ Scienc
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No